CLINICAL TRIAL: NCT05056857
Title: Neutrophil Functions in Breast Cancer
Brief Title: Neutrophil Extracellular Traps Formation in Breast Cancer Patients Taking Tamoxifen
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-0491; NCI-2021-09117 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0491 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical chart review): Patients undergo collection of blood samples and their medical charts are reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
  Other Names: Biological Sample Collection
Other: Electronic Health Record Review — Medical charts are reviewed

SUMMARY:
This study examines the long-term effects of tamoxifen (TAM) treatment on excessive production of neutrophil extracellular traps (NET) and their impact on breast cancer and side effects. NET are produced by the body to fight infections but have also been linked to side effects caused by the body's immune system. Treatment with tamoxifen increases the production of NETs. This study may help researchers determine if the increased number of NETs in the body has a damaging effect in breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the effect of long-term tamoxifen (TAM) treatment on excessive NET formation in breast cancer patients.

SECONDARY OBJECTIVES:

I. To understand the molecular mechanisms of tamoxifen-induced NET formation in breast cancer patients by examining the effect of long-term TAM treatment on the NET-induced factors.

II. To correlate the extend of NET formation with clinical data on tamoxifen resistance, drug side-effects, cancer metastasis and comorbidities.

EXPLORATORY OBJECTIVE:

I. To explore the association between the extent of NET formation and clinical data for breast cancer patients treated with TAM in combination with other drugs.

OUTLINE:

Patients undergo collection of blood samples and their medical charts are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age criteria for pre-menopausal group: Equal to or greater than 18 years of age and less than or equal to 45 years of age. Patients of age 46-50 will be included if they have not had menstrual cessation for 12 consecutive months.
* Age criteria for menopausal group: At least 51 years of age (median age of menopause). Menopause is defined as cessation of menstrual cycle for 12 consecutive months.
* Diagnosed with ER+ breast cancer
* Being treated with tamoxifen (TAM) for at least 6 months
* CONTROL SUBJECTS: Newly diagnosed ER+ breast cancer patients of the same age group as above on TAM for 0-6 months. This criterion is based on our preliminary results showing that patients taking TAM for 6-7 months exhibit near baseline level of NETs

Exclusion Criteria:

* Pregnant -The immune modulations geared toward maintenance of pregnancy are known to cause wide-spread alterations in innate and adaptive immune cell functions. In this scenario, divorcing the pregnancy-related changes in myeloid cell function from those relevant to sepsis and cancer will be complicated.
* History of severe congenital neutropenia due to genetic disorders, such as Kostmann Disorder (HAX1 gene mutation), ELA2 gene mutation, Wiskott-Aldrich syndrome (WAS), Growth Factor Independent 1 Protein (GFI1) gene mutation, Colony Stimulating Factor 3 Receptor (CSF3R) gene mutation, Schwachman-Diamond Syndrome, Barth Syndrome, WHIM Syndrome, and Chadiak-Higashi Syndrome (this list notably does not include Myelodysplastic Syndrome, or Acute/Chronic Myeloid Leukemia)
* History of autoimmune disorders, which can affect the body's inflammatory response, such as rheumatoid arthritis, lupus, Crohn's disease, multiple sclerosis, and psoriasis.
* History of chronic viral infections (human immunodeficiency virus [HIV], hepatitis), which can lead to reduced or variable immune cell function.
* A recent positive coronavirus disease (COVID) test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-menopausal and post-menopausal women diagnosed with estrogen receptor positive (ER+) breast cancer being treated with tamoxifen for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of neutrophil extracellular traps (NETs) in blood samples of pre- and postmenopausal women being treated with tamoxifen for varying periods of time. | through study completion, an average of 1 year
  Percent of NET-forming neutrophils is deduced in each sample by quantitative method standardized in the lab.

CONTACTS AND LOCATIONS:
Overall Officials: Jyotika Sharma, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org